CLINICAL TRIAL: NCT04567017
Title: Physical Activity of Staff on Medical Duty in a Department of Anesthesia and Critical Care During Guards
Acronym: AMAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO19103
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2019-09

CONDITIONS: Intensivist; Resident; Night Work
Keywords: Physical activity; guards; Intensive care
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
On-call work is an integral part of senior and junior patricians in a critical care department.

Several studies have examined the effect of sleep deprivation on physicians on call and the impact of sleep deprivation on the quality of patient care.

Some of these studies have shown that practitioners' concentration capacities have deteriorated as the guard progresses.

However, few studies have looked at the physical activity of practitioners over a period of on-call time (distance covered, number of steps,...), as well as other parameters than the time spent in communication over the telephone.

The age and seniority of practitioners seem to be factors that can influence these different parameters, and there are few figures in the literature.

DETAILED DESCRIPTION:
Practitioners and juniors will be informed of the study. If they agree to participate in the study, each volunteer will receive an assessment of their cognitive functions before taking up their duties via the Montréal Cognitive Assessment (MOCA) version 7.1.

The place of exercise (emergencies, anaesthesia and ICU Each participant will be equipped with a connected watch with pedometer and cardiofrequencemeter function (Fitness Tracker F07Max).

During his on-call period a questionnaire will be given to him, with socio-demographic data, sleep duration and quality and the number of acts during the on-call period.

The telephone data will be analysed by querying the internal telephone system of the Reims University Hospital.

At the end of the on-call period, the analysis of the data from the connected watch will be analyzed and each volunteer will benefit from an evaluation of his cognitive functions via the Montreal Cognitive Assessment (MOCA) version 7.3 after taking up his duties.

Data will be collected during 2 shifts for each practitioner and junior

ELIGIBILITY:
inclusion criteria :

- voluntary practitioners and residents of the critical care department (intensive care, emergencies and anaesthesia)

exclusion criteria :

* refusal to participate
* musculoskeletal disorders
* a significant medical history that prevents normal physical activity for age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: voluntary practitioners and residents of the critical care department (intensive care, emergencies and anaesthesia)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
measurement of physical activity in physician according to seniority | Day 1
  mean distance in meter according to seniority

SECONDARY OUTCOMES:
measurement of physical activity in physician | Day 1
  mean distance in meter
measurement of attention function | Day 1
  score in Birckenkamp D2-R test
sleep duration | Day 1
  average sleep time
quality of sleep | Day 1
  mean score on Spiegel scale

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France